CLINICAL TRIAL: NCT00489996
Title: A Multicenter, Randomized Trial Comparing a Combined Gemcitabine and Cisplatin 3-Week Regimen With a 4-Week Regimen in Non-Small Cell Lung Cancer Patients
Brief Title: Trial Comparing 3 and 4 Week Regimen of Gemcitabine and Cisplatin in Patients With Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6672; B9E-GH-JHSE
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gemcitabine
Drug: cisplatin

SUMMARY:
The purpose of this study is to evaluate response rate of the 3 week versus 4 week treatment of gemcitabine with cisplatin as the first line treatment for non-small cell lung cancer patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of NSCLC
* Presence of Stage IIIB or Stage IV disease
* Patients must have received no prior systemic chemotherapy
* Patients must have at least one bi-dimensionally measurable lesion with clearly defined margins and two perpendicular diameters that are clearly measurable by any of the following: chest x-ray, with at least one diameter 1.0 cm or greater, CT, with both diameters greater than the distance between cuts of the imaging study, palpation, with both diameters 2.0 cm or greater, or disease progressing in areas of prior radiation therapy may be included
* No prior radiotherapy for the target organ, no other radiotherapy for at least 2 weeks prior to study enrollment and the patient must have fully recovered from all acute toxic effects of the treatment.

Exclusion Criteria:

* Are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Are employed by Lilly (that is, employees, temporary contract workers, or designees responsible for the conduct the study). Immediate family of Lilly employees may participate in Lilly sponsored clinical trials, but are not permitted to participate at a Lilly facility. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have previously completed or withdrawn from this study or any other study investigating gemcitabine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-01; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Evaluate response rate

SECONDARY OUTCOMES:
Evaluate time to progression
Evaluate toxicities
Evaluate survival

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai, China

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com